CLINICAL TRIAL: NCT02208115
Title: A Comparison of the Appetite Responses to High and Low Glycemic Index Post-exercise Meals Under Matched Insulinemia and Fibre in Type 1 Diabetes
Brief Title: Post-exercise Appetite Responses in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: West-Walker3.1
Record Dates: First submitted 2014-07-25; First posted 2014-08-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; Exercise; Appetite
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Meal composition - High GI (Experimental): Changing the glycaemic index of the meal consumed after exercise (High GI versus Low GI).
  Interventions: Dietary Supplement: Meal composition - Low versus high GI.
- Meal composition - Low GI (Experimental): Changing the glycaemic index of the meal consumed after exercise (High GI versus Low GI).
  Interventions: Dietary Supplement: Meal composition - Low versus high GI.

INTERVENTIONS:
Dietary Supplement: Meal composition - Low versus high GI.

SUMMARY:
The investigators hypothesise that manipulating the glycaemic index of the meal after exercise will influence the acute appetite responses of Type 1 diabetes individuals

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-50 years old (male or female).
* Free from any diabetes related complications (apart from mild background diabetic retinopathy).
* HbA1c <8.5%.
* Not taking any prescribed medication other than insulin, and treated with a stable insulin regimen composed of a combination of slow/long acting insulin (glargine or detemir) and fast-acting insulin analogues (lispro or aspart), for a minimum of 6 months before the start of the study.
* Demonstrate normal cardiac function in response to exercise.

Exclusion Criteria:

* Aged younger than 18, or older than 50 years.
* Suffering from, or diagnosed with a diabetes related complication (apart from mild background diabetic retinopathy).
* HbA1c >8.5%.
* Currently taking prescribed medication, and not currently treated with a stable basal bolus regimen composed of a combination glargine or detemir, and lispro or aspart for at least 6 months before the start of the study.
* Failure to demonstrate normal cardiopulmonary responses during exercise, or have a medical condition which could prevent completion of exercise or be exacerbated because of.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Acute subjective appetite responses | 4 hours post-exercise
  Subjective appetite ratings via Visual Analogue Scales

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J West, PhD, Principal Investigator — Northumbria University
Locations (1):
- Clinical Research Facility, Royal Victoria Infirmary, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- [Derived] Campbell MD, Gonzalez JT, Rumbold PL, Walker M, Shaw JA, Stevenson EJ, West DJ. Comparison of appetite responses to high- and low-glycemic index postexercise meals under matched insulinemia and fiber in type 1 diabetes. Am J Clin Nutr. 2015 Mar;101(3):478-86. doi: 10.3945/ajcn.114.097162. Epub 2014 Dec 31. PMID 25733632